CLINICAL TRIAL: NCT04673500
Title: Comparison of Large Antecubital Vein Versus Small Vein on Dorsum of Hand for the Prevention of Propofol Injection Pain
Brief Title: Assessment of Pain on Propofol Injection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University Hospital (Other)
Responsible Party: Principal Investigator, Abdul Sattar Narejo, Consultant Anesthetist, King Khalid University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KingKhalidUH
Record Dates: First submitted 2016-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Injection Site Irritation
Keywords: Propofol; Injection pain; Veins

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two groups, eighty each. In all patients 15 to 30 minutes before shifting to the operation room a 20 gauge intravenous catheter was inserted either in a large antecubital vein (Group-1) or in a vein on dorsum of hand (Group-2). Lactate Ringer infusion was initiated at the rate of 120 ml/h. The arm was covered with green sheet. Patients received admixture of 2% lidocaine (1ml) in 1% propofol (19ml) either through large antecubital vein (Group-1, n = 80) or (Group-2, n = 80) through a vein at dorsum of hand. In both groups initially, thirty percent of the calculated dose of propofol (2mg/kg) was injected through an intravenous catheter. All patients were informed to report the researcher about the intensity of pain they experienced in numbers. Then induction of anesthesia was continued as routine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The whole arm with the intravenous catheter was covered with a green sheet, from where the mixture of propofol-lidocaine was given.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol-lidocaine through large vein (Experimental): Eighty patients randomly assigned in this arm received a 20 gauge intravenous catheter at the antecubital fossa and a mixture of 2% lidocaine 1 ml and 1% propofol 2mg/kg was given for induction of general anesthesia.
  Interventions: Drug: Propofol lidocaine through large vein
- Propofol-lidocaine through small vein (Placebo Comparator): Another eighty patients randomly assigned in this arm received a 20 gauge intravenous catheter at the dorsum of hand and a mixture of 2% lidocaine 1 ml and 1% propofol 2mg/kg was given for induction of general anesthesia.
  Interventions: Drug: Propofol lidocaine through small vein

INTERVENTIONS:
Drug: Propofol lidocaine through large vein — A mixture of 2% lidocaine 1 ml and 1% propofol 2mg/kg was given through a large antecubital vein to assess pain severity on propofol injection during general anesthesia induction
  Other Names: Group I
  Arms: Propofol-lidocaine through large vein
Drug: Propofol lidocaine through small vein — A mixture of 2% lidocaine 1 ml and 1% propofol 2mg/kg was given through a small vein on the dorsum of hand to assess pain severity on propofol injection during general anesthesia induction
  Other Names: Group II
  Arms: Propofol-lidocaine through small vein

SUMMARY:
Title: Assessment of pain on lidocaine-Propofol admixture injection: Comparing large antecubital vein and small vein dorsum of hand.

* Objective: To evaluate the pain on Propofol - lidocaine admixture injection using different sizes of veins on upper limb.
* Design: Prospective randomized clinical trial Place and duration of study: Department of Anesthesia, King Saud University Riyadh May 1, 2013 - May 31, 2014).
* Patient and methods: Total 160 adult patients were divided in two groups. Age 20-50 years of either gender, American Society of Anesthesiologist (ASA) class 1 and 2, scheduled for elective surgery under general anesthesia were included in the study. Patients with known history of allergy to lidocaine or Propofol, obese patients, anticipated difficult intubation, already on any analgesics and pregnant patients were excluded from the study. Both groups received an admixture of Propofol (1%) - lidocaine (2%) on induction of anesthesia through antecubital vein (Group- 1) or through a vein on dorsum of hand (Group- 2). Pain was assessed as none, mild, moderate or severe. Results: Moderate to severe pain on intravenous injection of Propofol-lidocaine admixture through antecubital vein and small vein on dorsum of hand was 20% vs 71%. Conclusion: There is marked reduction of pain when Propofol - lidocaine admixture was injected through antecubital vein as compared to small vein on dorsum of hand.
* Key words: Propofol, injection, pain

DETAILED DESCRIPTION:
Propofol is the most commonly used drug for induction of anesthesia because of its rapid onset, short duration of action, easy titration and with fewer hemodynamic Effects. Hypersensitivity reaction with Propofol is very rare and reported incidence of pain on injection is 26-70%. As Propofol is extensively used for the induction of anesthesia its pain on injection cannot be neglected. Propofol was launched for clinical practice in 1977 in Cremophor form and reformulation as aqueous solution was launched in 1986, an oil-in water emulsion containing soybean oil. Many interventions have been tried for the reduction of pain on Propofol aqueous solution injection. Unfortunately none of the intervention was found to be successful to abolish the pain completely. So far the mechanism of pain on Propofol injection is not clear.

The everyday uses of Propofol in many settings of the hospitals mandate its painless use. The proposed mechanisms of pain are release of local mediators and / or direct irritant effect of Propofol on nerve endings.

In this study the investigators combined two interventions, Propofol - lidocaine admixture and different size of veins, to evaluate the pain on Propofol injection. The admixture of Propofol-lidocaine was injected through two different sizes of veins which are commonly used for intravenous cannulations, large antecubital vein and small vein on dorsum of hand.

Propofol is a commonly used drug for induction of anesthesia and sedation in intensive care, emergency room and for endoscopic procedures. Unfortunately, despite its popularity pain on its injection is still unresolved problem. The exact mechanism of this pain is not clear so far.

Some investigators suggest that the lipid solvent for Propofol activates the plasma kallikrein-kinin system and produces bradykinin. This modifies the injected local vein causes vasodilation and hyper-permeability. This modification of the peripheral vein may increase the contact between the aqueous phase Propofol and free nerve endings of the vessel resulting in Pain.Others investigators believe that Propofol as a member of phenol group can have direct irritant effect on local vein by stimulating nociceptors and free nerve endings giving rise to an immediate sensation of pain. Based on these assumptions of Propofol induced pain pathway, different investigators postulated different interventions to alleviate this problem. Different pharmacological and non-pharmacological interventions have been tried for the reduction of pain on Propofol injection. The injection of Propofol through large antecubital vein was considered as a superior method than any other non pharmacology measures like changing the temperature of Propofol, large intravenous catheter and speed of injection.Pharmacological interventions with different drugs have been tried, pretreatment with lidocaine with venous occlusion. Propofol-lidocaine admixture, pretreatment with Ketamine, opioids,non-steroidal anti-inflammatory drugs ,magnesium sulfate, ondansetron, tramadol, acetaminophen, dexamethasone and Propofol emulsions containing medium and long chain triglycerides have been studied and reviewed extensively.

Among the all above interventions, Propofol lidocaine admixture is well known to be the best simple method. Lidocaine is a local anesthetic. It reduces the pain by two possible mechanisms, direct effect of local anesthetic on vascular smooth muscle and modifying the power of Hydrogen (pH) of Propofol. As lidocaine is a weak base solution when it dissolves with lipid it decrease the pH of the mixture. Thus, more Propofol in lipid phase cause less pain on injection.Injection of Propofol through large vein is another effective way in reducing pain. The vein diameter, flow rate, and endothelial structure might account for the reduction in pain. The injection of Propofol through a large antecubital vein, minimize the extent to which a high concentration of Propofol comes into contact with the sensitive endothelial wall. Furthermore Propofol will move faster from the injection site when more blood will be available to dissipate the bolus. Additionally, the composition of nociceptors along the endothelial wall might differ between the smaller veins of the hand and the larger antecubital veins. A meta-analysis showed that among the non-pharmacological and pharmacological interventions for the most effective method was the use of large antecubital vein followed by pretreatment with lidocaine combined with venous occlusion.

In this study the investigators have combined the two best and simple methods and compared the Propofol injection pain using two different sizes of veins on upper limb. The investigators have used small vein on dorsum of hand and large antecubital vein in the forearm. The investigators found that using large vein is superior to the small vein. Walker B.J. et al. reported that pretreatment with lidocaine using tourniquet is statistically superior to Propofol-lidocaine admixture. Whereas, Kim et al. investigated three doses of lidocaine mixed with Propofol 40 mg, 30 mg and 20 mg. The incidence of pain was 50%, 65% and 80% respectively.

In this study the investigators tested the efficacy of 20 milligram lidocaine in Propofol. When lidocaine -Propofol admixture was injected through small vein on dorsum of hand produces more pain as compared to large antecubital vein. This study results are comparable to the findings of Kim et al. However, combination of two strategies was unable to abolish Propofol injection pain completely. Based on these observations the investigators recommend whenever possible Propofol should be given in a mixture with lidocaine through large vein.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 50 years of either gender
* ASA ( American Society of Anesthesia) class 1 and 2
* Scheduled for elective surgical procedure under general anesthesia

Exclusion Criteria:

* Patients with known history of allergy to lidocaine or Propofol
* Obese patients
* Anticipated difficult intubation
* ASA 3 and 4
* Already on any analgesics and pregnant patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Assessment of severity of pain on propofol injection | From preoperative to day one postoperative
  A 20 gauge intravenous catheter was inserted either in large antecubital vein or in a small vein on dorsum of hand. An initial 30% of a mixture of propofol lidocaine was given to assess the severity of pain on propofol injection before the patient sleeps. The pain on propofol injection was assessed by numerical rating scale (NRS).
  0-10, where 0 is no pain and 10 is worst pain imaginable

SECONDARY OUTCOMES:
Heart rate | From base line pre-propofol injection to Intraoperative after full dose of propofol injection.
  Heart rate was assessed in association with pain on propofol injection

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Sattar Narejo, FCPS, FCAI, Principal Investigator — King Khalid University Hospital
Locations (1):
- Abdul Sattar Narejo, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marik PE. Propofol: therapeutic indications and side-effects. Curr Pharm Des. 2004;10(29):3639-49. doi: 10.2174/1381612043382846. PMID 15579060
- [Background] Sim JY, Lee SH, Park DY, Jung JA, Ki KH, Lee DH, Noh GJ. Pain on injection with microemulsion propofol. Br J Clin Pharmacol. 2009 Mar;67(3):316-25. doi: 10.1111/j.1365-2125.2008.03358.x. Epub 2008 Dec 10. PMID 19220277
- [Background] Dubey PK, Kumar A. Pain on injection of lipid-free propofol and propofol emulsion containing medium-chain triglyceride: a comparative study. Anesth Analg. 2005 Oct;101(4):1060-1062. doi: 10.1213/01.ane.0000166951.72702.05. PMID 16192520
- [Background] Nakane M, Iwama H. A potential mechanism of propofol-induced pain on injection based on studies using nafamostat mesilate. Br J Anaesth. 1999 Sep;83(3):397-404. doi: 10.1093/bja/83.3.397. PMID 10655909
- [Background] Ambesh SP, Dubey PK, Sinha PK. Ondansetron pretreatment to alleviate pain on propofol injection: a randomized, controlled, double-blinded study. Anesth Analg. 1999 Jul;89(1):197-9. doi: 10.1097/00000539-199907000-00035. PMID 10389803
- [Background] Jalota L, Kalira V, George E, Shi YY, Hornuss C, Radke O, Pace NL, Apfel CC; Perioperative Clinical Research Core. Prevention of pain on injection of propofol: systematic review and meta-analysis. BMJ. 2011 Mar 15;342:d1110. doi: 10.1136/bmj.d1110. PMID 21406529
- [Background] Walker BJ, Neal JM, Mulroy MF, Humsi JA, Bittner RC, McDonald SB. Lidocaine pretreatment with tourniquet versus lidocaine-propofol admixture for attenuating propofol injection pain: a randomized controlled trial. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):41-5. doi: 10.1097/AAP.0b013e31820306da. PMID 21455088
- [Background] Kim DH, Chae YJ, Chang HS, Kim JA, Joe HB. Intravenous lidocaine pretreatment with venous occlusion for reducing microemulsion propofol induced pain: comparison of three doses of lidocaine. J Int Med Res. 2014 Apr;42(2):368-75. doi: 10.1177/0300060513507391. Epub 2014 Mar 4. PMID 24595146
- [Background] Bano F, Zafar S, Sabbar S, Aftab S, Haider S, Sultan ST. Intravenous ketamine attenuates injection pain and arterial pressure changes during the induction of anesthesia with propofol: a comparison with lidocaine. J Coll Physicians Surg Pak. 2007 Jul;17(7):390-3. PMID 17686348
- [Background] Fujii Y, Itakura M. A comparison of pretreatment with fentanyl and lidocaine preceded by venous occlusion for reducing pain on injection of propofol: a prospective, randomized, double-blind, placebo-controlled study in adult Japanese surgical patients. Clin Ther. 2009 Oct;31(10):2107-12. doi: 10.1016/j.clinthera.2009.10.012. PMID 19922881 (Retraction: PMID 29724497 Clin Ther. 2018 Apr 30;:)
- [Background] Alipour M, Tabari M, Alipour M. Paracetamol, ondansetron, granisetron, magnesium sulfate and lidocaine and reduced propofol injection pain. Iran Red Crescent Med J. 2014 Mar;16(3):e16086. doi: 10.5812/ircmj.16086. Epub 2014 Mar 5. PMID 24829787
- [Background] Rahimzadeh P, Faiz SH, Nikoobakht N, Ghodrati MR. Which one is more efficient on propofol 2% injection pain? Magnesium sulfate or ondansetron: A randomized clinical trial. Adv Biomed Res. 2015 Feb 17;4:56. doi: 10.4103/2277-9175.151593. eCollection 2015. PMID 25802825
- [Background] Borazan H, Sahin O, Kececioglu A, Uluer MS, Et T, Otelcioglu S. Prevention of propofol injection pain in children: a comparison of pretreatment with tramadol and propofol-lidocaine mixture. Int J Med Sci. 2012;9(6):492-7. doi: 10.7150/ijms.4793. Epub 2012 Aug 15. PMID 22927775
- [Background] Canbay O, Celebi N, Arun O, Karagoz AH, Saricaoglu F, Ozgen S. Efficacy of intravenous acetaminophen and lidocaine on propofol injection pain. Br J Anaesth. 2008 Jan;100(1):95-8. doi: 10.1093/bja/aem301. Epub 2007 Oct 23. PMID 17959585
- [Background] Ahmad S, De Oliveira GS Jr, Fitzgerald PC, McCarthy RJ. The effect of intravenous dexamethasone and lidocaine on propofol-induced vascular pain: a randomized double-blinded placebo-controlled trial. Pain Res Treat. 2013;2013:734531. doi: 10.1155/2013/734531. Epub 2013 Jul 15. PMID 23956857